CLINICAL TRIAL: NCT05730647
Title: Prospective Observational Study of Adjuvant Hormone Treatment in Estrogen-receptor Positive Premenopausal Early Breast Cancer Patients
Acronym: GIM 23- POSTER
Status: Active, not recruiting | Type: Observational
Sponsor: Consorzio Oncotech (Other)
Responsible Party: Sponsor
Other Study IDs: GIM23-POSTER
Record Dates: First submitted 2023-02-07; First posted 2023-02-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Early Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: None intervention (observational study) — None intervention (observational study)

SUMMARY:
This will be a prospective, multicenter, observational study. The primary objective is to record the choice, in clinical practice, of adjuvant hormone therapy (tamoxifen, tamoxifen + LhRh, aromatase inhibitors + LhRh) in premenopausal patients with estrogen-receptor positive breast cancer.

The secondary objective is to correlate adjuvant hormone therapy choices with biological characteristics of the tumor (T size, lymph node status, grade, receptor level, Ki67, HER2 status) and patient characteristics (age, prior chemotherapy treatment).

ELIGIBILITY:
Inclusion Criteria:

1. - Premenopausal patients candidate to start adjuvant hormone therapy after breast cancer surgery
2. - Age >18 years
3. - No previous hormonal treatment
4. - Written informed consent

Exclusion Criteria:

1- Patient's inability to provide written informed consent 2 - Stage IV disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Premenopausal patients candidate to start adjuvant hormone therapy after breast cancer surgery.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2019-10-24 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2032-07-31 (Estimated)

PRIMARY OUTCOMES:
To record the choice, in clinical practice, of adjuvant hormone therapy. | 21 months
  Patients will be divided in groups according to type of adjuvant hormone therapy received:
  1. tamoxifen
  2. tamoxifen + LhRh
  3. aromatase inhibitor + LhRh Differences between groups will be evaluated with Chi-square test and Mann-Whitney test.

CONTACTS AND LOCATIONS:
Locations (40):
- Italy (40):
  - Centro di Riferimento Oncologico- IRCCS, Aviano
  - A.O. Consorziale Policlinico di Bari, Bari
  - IRCCS Istituto Oncologico di Bari, Bari
  - Osp. Papa Giovanni XXIII, Bergamo
  - Presidio Ospedaliero "Antonio Perrino" ASL Brindisi, Brindisi
  - Università degli Studi "G.d'Annunzio" Chieti-Pescara, Chieti
  - ASST Lariana - Ospedale S. Anna, Como
  - Azienda Ospedaliera S. Croce e Carle, Cuneo
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - I.R.C.C.S. A.O.U San Martino - IST, Genova
  - Ospedale Civile di Guastalla, Guastalla
  - Ospedale F.Renzetti di Lanciano, Lanciano
  - Ospedale S.M. Goretti, Latina
  - P.O. Vito Fazzi, Lecce
  - A.O. Ospedale Civile di Legnano, Legnano
  - AUSL Toscana Nord Ovest- Osp. Versilia, Lido di Camaiore
  - Ospedale di Macerata, Macerata
  - A.O.Papardo, Messina
  - A.O.U Policlinico di Modena, Modena
  - A.O.R.N. "A. Cardarelli", Napoli
  - AOU Federico II, Napoli
  - Azienda Ospedaliera Specialistica dei Colli - Ospedale Monaldi, Napoli
  - Istituto Nazionale dei Tumori - Fondazione G. Pascale, Napoli
  - Istituto Oncologico Veneto IRCCS, Padua
  - A. O. U. Pisana - Ospedale S. Chiara, Pisa
  - A.O.R. San Carlo, Potenza
  - Ospedale di Prato, Prato
  - AUSL della Romagna- P.O. di Ravenna, Lugo e Faenza, Ravenna
  - IRCCS Arcispedale S.Maria Nuova, Reggio Emilia
  - Fondazione Policlinico Gemelli, Roma
  - Istituto Nazionale Tumori Regina Elena, Roma
  - Ospedale San Camillo Forlanini, Roma
  - Policlinico Universitario Campus Biomedico, Roma
  - Istituto Clinico Humanitas Irccs, Rozzano
  - IRCCS Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Ospedale San Vincenzo, Taormina
  - Presidio Ospedaliero Martini - ASL TO1, Torino
  - Ospedale Santa Chiara, Trento
  - Azienda Ospedaliera Universitaria SM Misericordia, Udine
  - Ospedale San Pio da Pietrelcina, Vasto

IPD SHARING:
Plan to Share IPD: Undecided